CLINICAL TRIAL: NCT02970721
Title: Use of Psychotropic Medications Among Pregnant Women With Bipolar Disorder: Patterns, Determinants, and Impact on Perinatal Outcomes
Brief Title: Use of Psychotropic Medications Among Pregnant Women With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Kelly Anderson, Assistant Professor, Western University, Canada
Other Study IDs: 108217
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Bipolar Disorder; Pregnancy Complications
Keywords: bipolar disorder; adverse outcomes; readmission; polytherapy
MeSH Terms: conditions — Bipolar Disorder; Pregnancy Complications | interventions — Antipsychotic Agents; Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bipolar disorder-treated: Individuals in this group are taking any medication (mood stabilizer, antipsychotic, antidepressants, antianxiety) during pregnancy
  Interventions: Drug: Antipsychotic; Drug: Antidepressant; Drug: Antipsychotic and Antidepressant
- Bipolar Disorder-Not Treated: Individuals in this group are not taking any medications during pregnancy

INTERVENTIONS:
Drug: Antipsychotic — Antipsychotic monotherapy
  Groups: Bipolar disorder-treated
Drug: Antidepressant — Antidepressant monotherapy
  Groups: Bipolar disorder-treated
Drug: Antipsychotic and Antidepressant — Polytherapy
  Groups: Bipolar disorder-treated

SUMMARY:
The objectives of the proposed project are:

1. To describe the patterns of mood stabilizer, antipsychotic, antidepressant, and anxiolytic prescriptions during pregnancy over a period of 12 years (2002-2014) in women aged 13 to 50 years who are diagnosed with bipolar disorder in Ontario.
2. To identify the factors associated with use of antipsychotics, antidepressants, and antipsychotic-antidepressant polytherapy in pregnant women diagnosed with bipolar disorder.
3. To assess the impact of antipsychotics, antidepressants, and antipsychotic-antidepressant polytherapy on the risk of maternal, neonatal, and labour and delivery outcomes in women with bipolar disorder.
4. To assess the impact of antipsychotics, antidepressants, antipsychotic-antidepressant polytherapy on psychiatric readmission rates during the early postpartum period in women with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

Women were included in our study cohort if they met at least one of the following criteria: (i) an inpatient hospitalization with a primary discharge diagnosis of BD prior to the index pregnancy; (ii) an outpatient OHIP fee code for a mood disorder plus a prescription of a mood stabilizer prior to the index pregnancy (note that the outpatient OHIP fee code (296) without a prescription would not have been sufficient to identify BD patients because the fee code is used concurrently used for diagnosis of unipolar depression). Additionally, women were included in the study cohort if they were continuously covered for ODB throughout their pregnancy, defined as having filled any provincially funded drug prescription within six months prior to conception and another either during their pregnancy or within six months after delivery.

Exclusion Criteria:

(1) women with gestational weeks less than 20 and more than 45 at delivery; (2) pregnancies with multiple overlapping records over the study time period; (3) any data with inconsistencies and duplicate records for pregnancy; (4) any woman sharing the newborn's IKN, given that we would be unable to differentiate between the two persons; (5) observations with missing birth date for the baby and the time period between the mother's admission and discharge date greater than 14 days (since we were unable to determine the conception date for these women; and (6) women who filled a treatment prescription up to 30 days prior to pregnancy and none during the period of pregnancy.very

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women between the ages of 13 and 50 years who were hospitalized for a singleton obstetrical delivery between 2002-2014. Additionally, these women must be covered under the provincial drug benefit plan during index pregnancy, which is defined as having filled a drug prescription in the period from six months prior to pregnancy to six months after delivery. For women who had multiple pregnancies over the study period, we will select their first pregnancy as the index pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 3357 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maternal Outcomes (pregnancy) | 2002-2014
  Venous Thromboembolism, gestational diabetes, gestational hypertension, preeclampsia or eclampsia, placental abruption, placental infarction
Neonatal Outcomes | 2002-2014
  Preterm birth, small for gestational age, large for gestational age, sepsis, mortality, infection, neonatal adaption syndrome, respiratory distress syndrome, seizure, intraventricular haemorrhage
Fetal Outcomes | 2002-2014
  Stillbirth, congenital malformation
Labour and Delivery Outcomes | 2002-2014
  Caesarean, forceps/ventouse, induced labour, episiotomy or delivery with tear (3rd or 4th degree)
Psychiatric Readmission | 2002-2014
  Readmission for mental health reasons ≤ 7 days post-delivery, readmission for mental health reasons within 1 to 12 weeks post-delivery

REFERENCES:
- [Background] Boden R, Lundgren M, Brandt L, Reutfors J, Andersen M, Kieler H. Risks of adverse pregnancy and birth outcomes in women treated or not treated with mood stabilisers for bipolar disorder: population based cohort study. BMJ. 2012 Nov 8;345:e7085. doi: 10.1136/bmj.e7085. PMID 23137820
- [Background] Vigod SN, Gomes T, Wilton AS, Taylor VH, Ray JG. Antipsychotic drug use in pregnancy: high dimensional, propensity matched, population based cohort study. BMJ. 2015 May 13;350:h2298. doi: 10.1136/bmj.h2298. PMID 25972273
- [Background] Broeks SC, Thisted Horsdal H, Glejsted Ingstrup K, Gasse C. Psychopharmacological drug utilization patterns in pregnant women with bipolar disorder - A nationwide register-based study. J Affect Disord. 2017 Mar 1;210:158-165. doi: 10.1016/j.jad.2016.12.001. Epub 2016 Dec 8. PMID 28040641